CLINICAL TRIAL: NCT04972370
Title: Assessment of Secondary Cleft Lip and Nose Deformities in Patients With Repaired Unilateral Cleft Lip: A Proposal for a New Classification
Brief Title: A Proposal for a New Classification of Secondary Cleft Lip and Nose Deformities in Repaired Unilateral Cleft Lip
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Merna Labib Ebid-Allah, Plastic Surgery Resident, Sohag University
Other Study IDs: Soh-Med-21-07-08
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Patients With Unilateral Cleft Lip With or Without Cleft Palate
MeSH Terms: interventions — cyclopropapyrroloindole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Unilateral Cleft Lip with or without Cleft Palate
  Interventions: Other: Patients with Unilateral Cleft Lip with or without Cleft Palate

INTERVENTIONS:
Other: Patients with Unilateral Cleft Lip with or without Cleft Palate — 2 dimensional Photographs of patients with unilateral cleft lip with or without cleft palate

SUMMARY:
Congenital cleft lip with or without cleft palate is one of the most common congenital malformations with an estimated incidence of about 1 every 500 to 700 live births. Cleft lip and palate are caused by a complex combination of many environmental and genetic factors sharing into the etiology. Patients with cleft lip and palate undergo multiple surgeries to reconstruct the anatomy and function to achieve symmetric, aesthetic, and functional nasolabial region. The most important goals of correction of the cleft are to achieve an acceptable facial appearance and psychological and social well-being for the patient and his or her family. Therefore, assessment of nasolabial appearance following cleft surgery remains an important parameter for evaluating the outcome of the procedure. Unfortunately, some residual deformities in the nasolabial region such as the abnormal shape of the nose, scar of the upper lip, uneven white roll, notched or excess vermilion border will remain noticeable. So, the assessment of secondary cleft nasolabial deformities needs a reliable rating scale. Although many scoring systems have been described in the literature, there is no globally accepted reliable one. A frequently used scoring system is the one proposed by Asher-McDade that uses frontal and lateral view masked prints of the nasolabial area. The use of three-dimensional (3D) imaging seems to be the most reliable in assessing cleft-related facial deformities. However, scoring based on two-dimensional (2D) photographs is easier to perform and more applicable in daily practice because all cleft patients are photographed during their treatment journey at predetermined intervals. Assessment of secondary nasolabial deformities in cleft patients in large numbers of patients helps compare the aesthetic results of the different treatment protocols and techniques.

ELIGIBILITY:
Inclusion Criteria: All Patients with unilateral cleft lip who had undergone primary cleft lip repair surgeries during their first year of life at Sohag University Hospital from January 2006 to December 2020.

Exclusion Criteria:

1. Patients with multiple cleft lip repair surgeries.
2. If the primary cleft lip surgery was performed after the first year of life.
3. Patients with no available photographs

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with repaired unilateral cleft lip with or without cleft palate who had undergone primary cleft lip repair surgeries during their first year of life at Sohag University Hospital from January 2006 to December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Interrater reliability of a classification system that guides the need for secondary corrective surgery for patients with repaired unilateral cleft lip and having secondary cleft nasolabial deformities post-repair. | 6 months
  We compiled a photographic dataset of patients with secondary cleft nasolabial deformities post-repair. We developed a classification system of secondary deformities covering the key seven anatomical components, including nose, muscles, philtrum, lateral element, white roll, vermilion, and scar.
  Independent expert surgeons will evaluate each secondary deformity identified in the photographic dataset using a scoring system ranging from 0-2. 0 indicates acceptable secondary deformity, which requires no further surgery; 1 indicates secondary deformity that only requires corrective surgery upon patient parents' preference; 2 indicates significant secondary deformity requiring corrective surgery. We will measure the interrater reliability of the classification system. An agreement of 0.8 or more across the independent expert assessors will render the classification system valid for further prospective validation and clinical application.

REFERENCES:
- [Background] Mossey PA, Little J, Munger RG, Dixon MJ, Shaw WC. Cleft lip and palate. Lancet. 2009 Nov 21;374(9703):1773-85. doi: 10.1016/S0140-6736(09)60695-4. Epub 2009 Sep 9. PMID 19747722
- [Background] Dixon MJ, Marazita ML, Beaty TH, Murray JC. Cleft lip and palate: understanding genetic and environmental influences. Nat Rev Genet. 2011 Mar;12(3):167-78. doi: 10.1038/nrg2933. PMID 21331089
- [Background] Russell KA, Orthod D, Tompson B, Orthod D, Paedo D. Correlation between facial morphology and esthetics in patients with repaired complete unilateral cleft lip and palate. Cleft Palate Craniofac J. 2009 May;46(3):319-25. doi: 10.1597/07-143.1. Epub 2008 Sep 27. PMID 19642746